CLINICAL TRIAL: NCT02814253
Title: An Exploratory, Observational Clinical Evaluation of TidalSense's N-Tidal C Data-collector Capnometer to Collect Breathing Records in Patients With COPD
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Breathing Record Study
Acronym: CBRS
Status: Completed | Type: Observational
Sponsor: TidalSense (Industry)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: G001-15_CBRS
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Community Based Group: Patients who regularly present with exacerbations of COPD and have chronically-elevated CO2 levels. These patients are supported intensively in an out-patient setting (case-managed) and are potentially eligible for the community-based group.
- Acute Admissions Group: Patients who are admitted to hospital with an acute exacerbation of COPD. These patients are potentially eligible for the acute admission group.

SUMMARY:
This study is being done to collect information that will be used in the development of a new medical device. The new device is intended to help people with COPD to monitor their condition at home on a daily basis.

The device used in this study is called a capnometer. Different types of capnometer have been in use by doctors for many years. Capnometers measure the amount of carbon dioxide in your breath. The device that is used in this study is called the N Tidal C. It is a small, battery-powered personal device for you to use indoors either at home, at work or in hospital.

The study fits around the normal treatment, tests and medication of COPD patients and there will not be any changes made to the treatment of any study participants.

The study lasts for six weeks. Standard care clinical assessments will be taken at the start of the study, after 2 weeks, 4 weeks and 6 weeks. The tests for COPD include a check-up by the study doctor or nurse including the usual spirometry and blood gas tests. Each assessment visit will last for between 15-20 minutes.

At the start of the study each participant will be trained in the use of the device and they will be asked to use the device to record their normal relaxed breathing, 3 times a day (morning, afternoon and evening) every day for the 6- week period. A reading takes seventy-five seconds of ordinary breathing through the device.

Participants who feel unwell, or have an infection, will be asked to take more frequent breath records of up to six times a day if possible. This would be twice in the morning, twice in the afternoon and twice in the evening, leaving at least an hour between readings.

Participants will also be asked to complete a simple daily diary of how their health and COPD changes and information on the use of the device.

Participants will receive a telephone call 2 weeks after their last assessment visit to check how they are and to ask if any of their medicines have changed.

Participants will not benefit directly from taking part in this study and the device used in the study does not provide any feedback to them. The information we get from this study will help us to develop the device, and to learn more about the treatment and management of COPD.

DETAILED DESCRIPTION:
Study design: This is an uncontrolled, non-randomised, un-blinded longitudinal observational data collection study with the N-Tidal C data-collector capnometer in patients with COPD. Patients will be enrolled into one of two cohorts: community-based case managed patients with chronic hypercapnia, and hospitalised patients who have been admitted via the emergency room for the treatment of COPD-related ventilatory failure.

Patients who give informed consent will be screened for the study. Patients in the case-managed group will be screened at home or in routine clinic visits. Patients in the acute admission group will be screened after admission to hospital as soon as they are well enough to understand the study and to give written informed consent.

The N-Tidal C data-collector capnometer will be explained to the patients and they will be trained how to use it. Case-managed patients will be asked to use the device at home over a period of approximately 6 weeks, 3 times per day (morning, afternoon and evening), or 6 times per day if they feel that they are starting an infection or an exacerbation. Hospitalised patients will also use the device 3 times per day as in-patients and will then continue with the monitoring after discharge from hospital for a total period of 6 weeks. All patients will complete a daily diary record.

Case-managed patients will undergo clinical assessment of COPD during screening at home or in the COPD clinic; in-patients will undergo clinical assessment of COPD following admission and before discharge from hospital. All patients will be assessed a further 3 times: during the second and fourth week in the community, and at the end of the 6-week assessment period. A brief follow-up review will be conducted approximately 8 weeks after the start of capnometer monitoring. At each assessment, capnometry measurements will be taken in addition to routine spirometry, and arterial (in-patients) or capillary (in the community) blood gasses. The trial will not interfere with routine management of the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over.
* Diagnosed with moderate to severe COPD.
* Patients in the case managed group will have chronically elevated partial pressure of carbon dioxide (PaCO2) and be susceptible to frequent exacerbations of COPD.
* Patients in the acute admission group will have been admitted to hospital via the emergency room for treatment of COPD-related ventilatory failure .

Exclusion Criteria:

* Diagnosis of neuromuscular disorder.
* Diagnosis of Kyphoscoliosis.
* Patients who, in the opinion of the investigator, are unlikely to comply with the requirements of the study.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 30 men and women with a diagnosis of moderate to severe COPD.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To collect a longitudinal observational study database of capnograph records for up to 30 patients with COPD using the N-Tidal C data-collector capnometer. | 4 months

SECONDARY OUTCOMES:
To identify the correlation of carbon dioxide (CO2) measurements by capnography with those obtained by periodic standard arterial and capillary blood gas measurements. | 12-18 months
To identify the within-day and day-to-day variability of exhaled carbon dioxide in patients with COPD. | 12-18 months
To measure the absolute change in exhaled carbon dioxide measurements of patients admitted with an acute exacerbation of COPD during their recovery. | 12-18 months
To capture the carbon dioxide signature predictive of exacerbation in monitored patients who undergo an acute admission during the study. | 12-18 months

OTHER OUTCOMES:
To assess the ability of patients with COPD to use the N-Tidal C data-collector capnometer daily and to capture user feedback. | 12-18 months
To assess the frequency of replacement of the consumable mouthpieces and batteries in normal daily use. | 12-18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Mahadeva, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Derived] Talker L, Neville D, Wiffen L, Selim AB, Haines M, Carter JC, Broomfield H, Lim RH, Lambert G; BRS Study Team; Weiss ST, Hayward G, Brown T, Chauhan A, Patel AX. Machine diagnosis of chronic obstructive pulmonary disease using a novel fast-response capnometer. Respir Res. 2023 Jun 2;24(1):150. doi: 10.1186/s12931-023-02460-z. PMID 37268935